CLINICAL TRIAL: NCT05062499
Title: The Effects of Home Use of Transcutaneous Electrical Nerve Stimulation on People With Knee Osteoarthritis (OA) and or Chronic Knee Pain
Brief Title: The Effects of Home Use of Transcutaneous Electrical Nerve Stimulation on People With Knee OA and or Chronic Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDV-CDD-210023
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Knee Pain Chronic; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS (Active Comparator): electrical stimulation
  Interventions: Device: Active TENS
- Sham TENS (Sham Comparator): no stimulation
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: Active TENS — electrical stimulation
  Arms: Active TENS
Device: Sham TENS — no stimulation
  Arms: Sham TENS

SUMMARY:
The purpose of the research is to see if the use of transcutaneous electrical nerve stimulation (TENS) at home would reduce knee pain and swelling in people with knee OA and/or chronic knee pain.

ELIGIBILITY:
Inclusion Criteria:

* The inclusionary criteria for subjects: Male or Female with the age of 45 years or older, ultrasonography scale of 0-3 for grading of primary Knee OA of the knees, pain perceived as a minimum of 3/10 and a maximum of 7/10 weekly average during the baseline period on a 0-10 active VAS pain scale, no phobia of electrical stimulation, no pain or anti-inflammatory medication will be taken during the study. Injury/pain that began at the knee a minimum of 6-weeks before entering the study.

Exclusion Criteria:

* Exclusion criteria for the subjects: Pregnancy, Diabetes Mellitus, Neuropathy, Smoker, Uncontrolled HTN, Past surgery in the region to be treated by TENS or had received an intra-articular corticosteroid or hyaluronic acid injection within 6 months before enrollment, Arthritis (RA) in the area to be treated by TENS, Allergic to tape/electrodes, Dementia, history of knee joint replacement or tibial osteotomy, undergoing physical therapy, any other major joint pain (e.g., back, hip, or ankle) that could limit functional ability, contraindications to TENS (pacemakers, dermatological conditions, and abnormal sensation in the knees), severe medical or neurological conditions (e.g. Chronic obstructive pulmonary disease, cardiovascular disease, arteriosclerosis obliterans, cerebrovascular accident, lumbar disc, herniation, and rheumatoid arthritis) or do not utilize stairs in daily living and unable to walk without ambulatory assistive devices. The candidate will be disqualified as a subject for the study if less than 5 days of pedometer use or less than 5 days VAS reporting within the prior week's baseline period.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Knee pain evaluated using the VAS for the stair climb test. | 10min
  The mean knee pain during the stair climb test is timed up and go test, and the 6-minute walk test will be measured using the VAS. Participants will record their level of knee pain by drawing a vertical mark between the ends of a 10-cm horizontal line. The 0-cm end and the 10-cm end represented no pain and the most extreme pain, respectively. The distance from the 0-cm end to the drawn mark was recorded to the first decimal place.
6-minute walk test (6MWT) | 15min
  In the 6-minute walk test, the participants will walk as far as they could within 6 minutes. They will be not allowed to carry a watch or provided feedback during the trial. Although rest periods are allowed, time recording will continue. The participants will be encouraged at 1-minute intervals. Their performance will be measured as the total distance traveled, and be recorded as an integral number.
Timed Up and Go (TUG) test | 10min
  The participant will sit down at first and then stand up when given the signal to start. As fast as possible, the participant will walk 3 meters toward a cone on the floor, circle it, walk back 3 more meters toward a chair, and finally sat sit down. Timing begins on the signal to start and ends when the participant completely sits down with their back resting on the backrest of the chair. Two trials will be performed, and the faster time of the 2 trials will be recorded to the nearest one-hundredth of a second.

SECONDARY OUTCOMES:
knee extensor strength | 10min
  The maximum isometric knee extensor strengths will be measured using a handheld dynamometer (HHD), which is the validated method in previous research on elderly individuals who are prone to falls.15 The maximum force will be recorded in Newtons (N), and testing will be repeated for 2 measurements. The averaged value of 2 measurements was used for statistical analysis.